CLINICAL TRIAL: NCT01678599
Title: Optimization of Sampling Procedure for PCR Technique to Assess Parasitological Response for Patients With Chronic Chagas Disease Treated With Benznidazole in Aiquile, Bolivia
Brief Title: Optimization of PCR Technique to Assess Parasitological Response for Patients With Chronic Chagas Disease
Acronym: PCR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSF/DNDi-CD-PCR-01
Record Dates: First submitted 2012-03-01; First posted 2012-09-05 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Chagas Disease
Keywords: Chagas Disease; PCR; diagnosis
MeSH Terms: conditions — Chagas Disease; Disease | interventions — benzonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benznidazol (Other): This is a single arm, open label study; therefore, all subjects enrolled will receive benznidazol.
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: Benznidazole — All patients participating in this study will be treated with Benznidazole, 5mg/Kg/day PO BID for 60 days with a maximum daily dose of 300mg, as per routine care provided by MSF in rural communities in Aiquile. For patients > 60 kg, the total dose should be calculated (5mg/Kg x Weight x 60 days) and treatment duration should be adjusted/prolonged accordingly. This treatment is in accordance with the local recommendations from the Ministerio de Salud y Deportes de Bolivia.
  Other Names: LAFEPE Benznidazol

SUMMARY:
The purpose of this study is to estimate the gain in sensitivity of several multiple-sample strategies of PCR samples with respect to the current standard (single sample of 10 ml) to detect Chagas chronic stage at baseline and to identify the optimal sampling strategy based on the sensitivity, cost,the completeness of sampling and the acceptability for study patients.

DETAILED DESCRIPTION:
Chagas Disease (CD) ranks among the world's most neglected diseases. In Latin America, 21 countries are endemic for CD with an estimated 108 million people at risk of contracting the disease. Estimates from the 1980s indicated that some 16 -18 million individuals were infected. In the 1990s, after a series of multinational control initiatives, estimates of the number of infected people were revised to 9.8 million in 2001. The estimated burden of disease in terms of disability-adjusted life years (DALYs) declined from 2.7 million in 1990 to 586,000 in 2001. Recent estimates from Pan-American Health Organization (PAHO), 2006 indicate 7.54 million infected people and 55,185 new cases per year. CD,also known as American trypanosomiasis,is a zoonotic disease caused by the protozoan hemoflagellate Trypanosoma cruzi that is mainly transmitted by large, blood-sucking, reduviid bugs of the subfamily Triatominae. Clinically, human CD has two phases, acute and chronic. The acute phase, which lasts a few weeks, is a febrile and toxemic illness, during which the parasite can be detected by direct examination of fresh blood. In the chronic phase, the diagnosis depends on hemocultures of varying degree of sensitivities, xenodiagnosis, PCR or detecting IgG antibodies. Untreated, the chronic phase continues for the rest of a person's life. It begins with no specific symptoms or clinical manifestations for a period of approximately 10 or 15 years, the "indeterminate form" of the disease. About 20 to 50% of chronic Chagas patients over the ensuing years, depending on the endemic area analyzed, will develop involvement of the heart or gastrointestinal tract. Current therapy for CD is limited to two nitroheterocyclic drugs, Nifurtimox and Benznidazole, the later being the most widely used drug for Chagas disease treatment. The indications for treatment are acute disease (including congenital infection), and early chronic disease (that is, in children < 15 years of age and patients in the early phase of chronic infection), plus reactivation of the infection by immunosuppression.

Late chronic phase is treated at the clinician's discretion. In a hierarchy of need, it has been argued that patients in the indeterminate phase of the disease would represent the main target population for evaluation of new treatments. With decreasing incidence of the disease, even in countries with the highest number of new cases, the highest disease burden is among patients in the asymptomatic, chronic phase of the disease. Bolivia, for example, has at least 200,000 children under the age of 15 years and 1 million adults infected with T. cruzi, for an estimated total of 700,000 people with the indeterminate form or asymptomatic, chronic phase. The development of effective and affordable treatment for the millions of people with ongoing infections and the prevention of chronic complications is recognized as a key disease control priority in CD. The evaluation of cure is considered the most complex aspect of treatment in CD, leading to often diverse and controversial results. The term parasitological cure is of difficult interpretation and the evaluation challenging, in light of the need for total elimination of parasites not only from blood but also from tissue. Clinical cure demands long-term evaluation and is often of uncertain nature due to the pathogenesis of the disease, with the action of the parasite, the host response and their consequent clinical manifestations evolving for long period of times. Over recent years an increasing body of data has pointed to a strong biological rationale for the use of parasitological outcomes as surrogate markers for acute and indeterminate Chagas disease. There is increasing evidence of the role of T. cruzi persistence in the perpetuation of immune response and evolution of the disease. Also, recent non-randomized clinical trials with long-term follow-up have demonstrated a positive effect from anti-parasitic chemotherapy in patients with chronic CD and the correlation of these findings with serology results. Therefore, for the purposes of clinical development and proof-of-concept, it has been suggested that parasitological and serological tests be used for the assessment of response in both acute and chronic disease. A negative direct smear at the end of treatment is generally accepted as evidence of response in acute patients. In chronic disease, serial hemoculture, xenodiagnosis or PCR can be used to support serological assessment and a positive parasitological result indicates treatment failure. Hemoculture and xenodiagnosis are techniques that may present low sensitivity in chronic patients, they require proper resources/infrastructure and very skilful personnel. In regards to conventional serology, with indeterminate chronic patients, a decrease in antibody titers may take up to 5 years with seroconversion to negative occurring after 5-10 years. In consequence, it is proposed that efficacy assessment for clinical studies in indeterminate disease be done with the use of qualitative and quantitative PCR. However, there has been significant variability in the clinical sensitivity and specificity of PCR in published studies, with differences seen across phases of the disease and a number of techniques in use requiring standardization. In particular, there has been concern regarding the sensitivity of PCR in chronic Chagas disease due to the low levels of circulating parasites and natural fluctuations of the parasitaemia. Latest studies have shown a broad dynamic range for PCR use allowing direct measurements in cases with high parasitic loads such as immunosuppressed Chagas disease patients and congenitally infected newborns, as well as in cases with low parasitaemias, such as patients at the indeterminate phase or under etiological treatment. PCR testing has also been used for early detection of T. cruzi reactivation after heart transplantation, with documented detection of parasitic load increase, previous to diagnosis of clinical reactivation. In addition, there are accruing clinical and experimental data suggesting a degree of correlation between parasitaemia and tissue infection. Another important advance in recent years has been the TDR sponsored-study for standardization and laboratory validation of qualitative PCR testing for T. cruzi. Standardized procedures for qualitative assessment of PCR (standard and real-time PCR) yielding higher analytical sensitivity and specificity, reproducibility, with low levels of intra- and inter-assay variation and accuracy have been selected. Results from this exercise have been presented in a meeting in Buenos Aires, Nov 08, and they are expected to be published in the near future. However, there is limited information on the efficacy of treatment for chronic indeterminate CD patients, and only a few studies employed PCR to assess parasitological response. A panel of experts in CD at three meetings hosted by DNDi and the CD protocol development team gave support to the evaluation of PCR as a marker for parasitological response in indeterminate chronic disease. During these discussions,there was consensus on the value of using serial blood collections for qualitative PCR assays in order to increase PCR testing sensitivity.

Data in support of this information are limited to an Argentinean cohort of 41 pregnant women followed-up with monthly blood collections. In this small group, PCR sensitivity was 60,2% for a single collection, 74% for 2 blood collections and 80,5% for 3 blood collections (A. Schijman, manuscript in preparation). In addition, a study from Castro published in 2002 indicated a significant increase from 70.0% to 81.7% in the sensitivity of PCR with the addition of a second sample (P=0.03). The addition of a third sample led to non-significant increase in sensitivity to 86.7%. Unfortunately, the sample size was small, there was no indication of the interval of sampling and the qualitative PCR technique was non-standardised. During the panel discussions, there was no agreement on the precise interval for serial sampling, in view of the lack of information in support for a definite interval for blood sampling to maximize sensitivity. Data obtained with xenodiagnosis suggest the absence of both circadian rhythm and T. cruzi periodicity with in chronic chagasic individuals. Therefore, when defining sampling procedures, one would need to balance the gain on the PCR sensitivity and logistics/feasibility in conducting clinical trials in a field setting. In order to prepare for future clinical trials on CD, DNDi acknowledges the need to evaluate and optimize the procedures for PCR implementation as a tool of parasitological assessment in patients with chronic indeterminate form of CD. Study ethical approval will be sought from the Médecins Sans Frontières Ethical Review Board and, the Ethical Review Board from the Colectivo de Estudios Aplicados y Desarollo Social (CEADES), Cochabamba, Bolivia. Furthermore, the study will be submitted and reviewed by the National Chagas Control Program and the 'Comité de Ética e Investigación' del Ministerio de Salud, Bolivia. This is a descriptive study aiming to assess whether multiple PCR blood sampling procedures at baseline can provide higher sensitivity compared to single sampling, as well as their feasibility in a field setting. Blood sampling for baseline and EOT will be as follows: one initial blood sample of 10 mL (Sample 1), followed by 1 blood sample of 5mL collected immediately following (Sample 2); plus one blood sample of 10mL collected 1 week later (Sample 3). Total of 3 blood samples. At the 6 and 12 months follow-up visits, only the optimal sampling strategy at EOT will be used.

Sampling strategies:

In order to explore PCR sensitivity according to the number of blood samples, PCR results will be analyzed as single assays as well as, at the data analysis stage, by combining PCR results for patients at a given time-point.

* Reference to be used Current strategy (CS): Sample 1 : Single sample of 10 ml Two major types of strategies may be developed and need an assessment:
* Reinforcement Strategy (RS) that consists in adding blood sampling(s) to the current single-sample approach (volume of 10 ml). Unless additional samplings do not allow the detection of additional PCR-positive cases (which is unlikely) such strategy will inevitably be more sensitive than the current one.
* Substitution Strategy (SS) that consists in replacing the current approach (sample 1 = 10 ml) by a 5 ml sampling (sample 2) and possibly further sampling(s) (sample 3). These strategies are not necessarily better than the current one.

Study Site:

The present study will be conducted in rural communities in the municipalities of Aiquile, Omereque and Pasorapa in the province of Narciso Campero, Bolivia, where Médecins Sans Frontières has established a program for "Chagas disease prevention, diagnosis and treatment" in partnership with the local health authorities. The local population is ~ 40,000 individuals, living in one of the areas with highest burden of CD in the country. In the context of this program, the individuals living in rural communities will be screened for Chagas disease and those who fulfil eligibility will be invited to participate in the study. Equal opportunities for treatment and management of the disease will be provided by MSF and its partners to all Chagas positive subjects, despite participation or not in the study.

Main Entry Criteria:

Inclusion / Exclusion Patients with chronic CD that have the indication for treatment with benznidazole. Patients must fulfil the following eligibility criteria for enrolment in the study:

Inclusion criteria:

* Age between > 18 - 60 years
* Diagnosis of T. cruzi infection by Chagas serology. Two out of three serological tests must be positive (conventional ELISA, recombinant ELISA, or HAI)
* Written informed consent form

Exclusion criteria:

* Women in reproductive age who have a positive pregnancy test at screening, or who are breastfeeding Note: Women in reproductive age must accept to use a contraceptive method during the entire treatment phase of the trial
* Current presentation of serious health condition such as: active pulmonary tuberculosis and clinical signs of liver or renal failure.
* Chagas cardiomyopathy stage II, III and IV (according to the NYHA classification)
* Subjects requiring pacemaker implantation or other serious cardiac conduction defects
* History of CD treatment with benznidazole or nifurtimox at any time in the past
* Inability to comply with follow-up and/or not having a permanent address
* History of alcohol abuse or any other drug addiction Note: all patients participating in this study will be treated with Benznidazole, 5mg/Kg/day PO BID for 60 days, as per routine care provided by MSF in rural communities in Aiquile. This treatment is in accordance with the local recommendations from the Ministerio de Salud y Deportes de Bolivia. The participation of the patient in this study is voluntary and his refusal or withdrawal of consent at any time during the study will not affect his/her right to receive treatment for Chagas disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between > 18 - 60 years
* Diagnosis of T. cruzi infection by Chagas serology. Two out of three serological tests must be positive [conventional ELISA, recombinant ELISA, or HAI)
* Written informed consent form

Exclusion Criteria:

* Women in reproductive age who have a positive pregnancy test at screening, or who are breastfeeding Note: Women in reproductive age must accept to use a contraceptive method during the entire treatment phase of the trial
* Current presentation of serious health condition such as: active pulmonary tuberculosis and clinical signs of liver or renal failure.
* Chagasic cardiomyopathy stage II, III and IV (according to the NYHA classification)
* Subjects requiring pacemaker implantation or other serious cardiac conduction defects
* History of CD treatment with benznidazole or nifurtimox at any time in the past
* Inability to comply with follow-up and/or not having a permanent address
* History of alcohol abuse or any other drug addiction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are: - A positive or negative PCR at baseline (BL) among serology positive patients. | Bloods will be at baseline and EOT (last day of treatment +10 + 5 days), 6 months and 12 months follow-up visits.
- Identification of the optimal relationship between sensitivity and feasibility at baseline. | Bloods will be at baseline and EOT (last day of treatment +10 + 5 days), 6 months and 12 months follow-up visits.
  For BL and EOT visits, blood samples will be as follows: one initial blood of 10 mL (Sample 1), followed by 1 sample of 5mL collected immediately following (Sample 2); plus one blood sample of 10mL collected 1 week later (Sample 3).
  Once the optimal strategy has been defined for EOT visit (see section 10.7), this will be the strategy of blood collection to be used at the 6 and 12 months follow-up visits

SECONDARY OUTCOMES:
- Identification of the optimal relationship between sensitivity and Identification of the optimal relationship between sensitivity and feasibility at End Of Treatment (EOT) | Bloods will be at baseline and EOT (last day of treatment +10 + 5 days), 6 months and 12 months follow-up visits.
- The proportion of patients who convert from PCR (+) at baseline to PCR (-) at EOT - to be estimated using 1) the current sampling schedule (CS), the most sensitive one and the optimal one. | Bloods will be at baseline and EOT (last day of treatment +10 + 5 days), 6 months and 12 months follow-up visits.
- The proportion of patients who convert from PCR (+) at baseline to PCR (-) at 6 and 12 months follow-up - to be estimated using 1) the current sampling schedule (CS) and the optimal one (based on EOT data). | Bloods will be at baseline and EOT (last day of treatment +10 + 5 days), 6 months and 12 months follow-up visits.
- Relative reduction [(parasite count at baseline - parasite count at EOT, 6 and 12 months)/parasite count at baseline] of parasitemia - to be evaluated through parasite load at EOT, 6 and 12 months through quantitative PCR. | Bloods will be at baseline and EOT (last day of treatment +10 + 5 days), 6 months and 12 months follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Loza, Biochemist, Principal Investigator — Medicin Sans Frontièrs
Locations (1):
- Medicin Sans Frontièrs (MSF), Aiquile, Bolivia

REFERENCES:
- [Background] Duffy T, Bisio M, Altcheh J, Burgos JM, Diez M, Levin MJ, Favaloro RR, Freilij H, Schijman AG. Accurate real-time PCR strategy for monitoring bloodstream parasitic loads in chagas disease patients. PLoS Negl Trop Dis. 2009;3(4):e419. doi: 10.1371/journal.pntd.0000419. Epub 2009 Apr 21. PMID 19381287
- [Derived] Parrado R, Ramirez JC, de la Barra A, Alonso-Vega C, Juiz N, Ortiz L, Illanes D, Torrico F, Gascon J, Alves F, Flevaud L, Garcia L, Schijman AG, Ribeiro I. Usefulness of Serial Blood Sampling and PCR Replicates for Treatment Monitoring of Patients with Chronic Chagas Disease. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01191-18. doi: 10.1128/AAC.01191-18. Print 2019 Feb. PMID 30509941
- See also: Drugs for Neglected Diseases initiative — http://dndi.org